CLINICAL TRIAL: NCT00947570
Title: Neural Substrates of Anticipation and Interoception in Anxiety Disorders
Brief Title: Neural Functioning Underlying Anxiety and Its Treatment (The INSULA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Murray B. Stein, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01MH065413 (NIH); R01MH065413 (NIH); DATR A2-AIA
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorders
Keywords: Cognitive Behavioral Therapy; Functional Brain Imaging; Psychotherapy; Treatment; Brain Imaging
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive behavioral therapy (Experimental): Participants with panic disorder or generalized anxiety disorder (GAD) will receive a course of individual cognitive behavioral therapy targeted at their principal disorder.
  Interventions: Behavioral: Cognitive behavioral therapy for anxiety

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for anxiety — 10 sessions delivered over the course of 14 weeks and aimed at reducing pathological behaviors and patterns of thought
  Other Names: CBT; Behavior Therapy

SUMMARY:
This study will examine the effects of cognitive behavioral therapy on brain function in people with anxiety disorders.

DETAILED DESCRIPTION:
Anxiety disorders are characterized by excessive and irrational fears of common situations that impair normal functioning. Neuroimaging allows researchers to examine brain functioning as people are presented with tasks that provoke or model anxiety. Neuroimaging research suggests that anxiety is moderated by a neural circuit involving three parts of the brain: the amygdala, the insula, and the prefrontal cortex (PFC). Increased activation of the amygdala and insula is associated with high anxiety, although activation of the PFC is thought to reduce anxiety. Cognitive behavioral therapy (CBT) is the only type of psychotherapy with strong evidence for effectively treating panic disorder (PD) and generalized anxiety disorder (GAD), but it only works about half the time. This study will use neuroimaging to examine when and how CBT affects brain functioning in people with PD and GAD. The long-term goals of the research are to develop neuroimaging as a diagnostic tool, to use neuroimaging to predict treatment response, and to understand which changes in brain functioning are related to successful treatment.

Participation in this study will last approximately 3 months. Four groups of participants will be recruited: healthy controls and people with PD, GAD, or social phobia (SP). All participants will undergo functional magnetic resonance imaging (fMRI) scanning-a measure of brain functioning-at the first visit. During the fMRI scan, participants will be asked to perform computerized tasks that involve responding to images. This will be the only visit that the healthy controls and people with SP complete; their inclusion in the study establishes a comparison point for the brain scans of the other participants. People with PD and GAD will then be asked to complete 10 sessions of CBT over a 10- to 14-week period. After 3 months, these participants will again undergo fMRI scanning. At 3 and 6 months after the completion of CBT, these participants will be asked to complete follow-up questionnaires about their anxiety.

ELIGIBILITY:
Inclusion Criteria:

* High school or higher education
* DSM-IV diagnosis of panic disorder (with ongoing symptoms), generalized anxiety disorder, or both

Exclusion Criteria:

* Lifetime diagnosis of psychotic disorder, organic mental disorder, or bipolar I disorder
* Substance dependence within the last 12 months or diagnosis of alcohol or substance abuse within the past month
* Use of psychotropic or anti-epileptic medications within the past 6 weeks
* Heavy caffeine use, defined as drinking more than 6 caffeinated beverages per day
* Current smoker
* Possibility of pregnancy
* History of claustrophobia or difficulty lying flat for long periods
* Ferrous metal in the body

Exclusion Criteria for Healthy Controls only:

* Lifetime diagnosis of major depressive disorder (MDD), bipolar I or II disorder, panic disorder (PD), agoraphobia without panic, generalized anxiety disorder (GAD), social phobia (SP), post-traumatic stress disorder (PTSD), obsessive-compulsive disorder (OCD), or an eating disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) response in amygdala, insula, and medial prefrontal cortex, as measured with functional magnetic resonance imaging (fMRI) | Measured at baseline and after 10 to 14 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Murray B. Stein, MD, MPH, Principal Investigator — University of California, San Diego

REFERENCES:
- See also: Click here for more information on the UCSD Anxiety Disorders Research Program — http://www.veryshy.org/research/